CLINICAL TRIAL: NCT02708134
Title: Quality of Pediatric Resuscitation in a Multicenter Collaborative: An Observational Study
Brief Title: Quality of Pediatric Resuscitation in a Multicenter Collaborative
Acronym: pediRES-Q
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-012099
Record Dates: First submitted 2016-01-28; First posted 2016-03-15 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest
Keywords: Chest compressions; Cardiopulmonary Resuscitation; Pediatric
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Cardiac Arrests: Pediatric cardiac arrests requiring chest compressions for at least 1 minute managed at clinical centers identified as part of standard clinical operations.

SUMMARY:
This is a prospective, observational, multi-center cohort study of pediatric cardiac arrests.

The purpose of the study is to determine the association between chest compression mechanics (rate, depth, flow fraction, compression release) and patient outcomes. In addition, the investigators will determine the association of post cardiac arrest care with patient outcomes.

DETAILED DESCRIPTION:
Cardiac arrests in children are a major public health problem. Thousands of children each year in the USA are treated with cardiopulmonary resuscitation (CPR) and managed after their cardiac arrest. Neurological outcomes following these in-hospital CPR events are often abnormal. As children with neurological deficits following CPR are a major burden for families and society, improving neurological outcomes through superior chest compression delivery during CPR and optimal care and management after cardiac arrest is an important clinical goal.

Therefore, the objective of this investigation is to obtain evidentiary support to associate the relationship of quantitative CPR quality data (depth, rate, chest compressions (CC) fraction, compression release) during CPR, post-cardiac arrest care (PCAC) and patient survival in those children who suffer an arrest within the study (RES-Q) Network.

ELIGIBILITY:
Inclusion Criteria:

* Patient received chest compressions for at least 1 minute
* Patient between gestational age ≥37 weeks and 18 years of age

Exclusion Criteria:

* Patient on veno-arterial extracorporeal membrane oxygenation (ECMO) therapy at beginning of CPR event

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Data will be collected from pediatric cardiac arrest events as part of standard clinical operations.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Aggregate score composed of American Heart Association (AHA) recommended depth, rate, and chest compression fraction during CPR | 10 Years
  Primary outcome: "Guideline-compliant CPR" which will be determined by an aggregate score comprised of the following three components: depth, rate, and chest compression fraction. The three components will be analyzed in 30 and 60 second epochs. "Guideline-compliant CPR" requires that each component meet the following criteria: 1) Age-determined American Heart Association (AHA) guideline recommended depth; 2) rate ≥ 90 and ≤ 120 CC/min; and 3) CC Fraction ≥ 0.80. Depth, rate, and CC Fraction will be calculated for each epoch and an aggregate score will be assigned. The primary analysis will be performed on that total score.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (61):
- United States (40):
  - Kaiser Permanente, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Chldren's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Wilmington, Delaware
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Lurie Children's (Children's Hospital of Chicago), Chicago, Illinois
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Kentucky Children's Hospital, Lexington, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Mount Sinai Kravis Children's Hospital, New York, New York
  - Morgan Stanley Children's Hospital, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Upstate Golisano Children's Hospital, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Akron Children's, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center, Austin, Texas
  - Medical City Children's Hospital, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Perth Children's Hospital, Nedlands
  - Queensland Children's Hospital, South Brisbane
- Sabara Hospital Infantil, São Paulo, Brazil
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's, Vancouver, British Columbia
  - Alberta Children's, Calgary
- Instituto Roosevelt, Bogotá, Colombia
- IRCCS Ospedale Pediatrico Bambino Gesù, Roma, Italy
- Japan (3):
  - Aichi Children's Health and Medical Center, Aichi
  - Kobe Children's Hospital (Hyogo Prefectural), Kobe
  - Tokyo Metropolitan Children's Medical Center, Tokyo
- Erasmus MC - Sophia Children's, Rotterdam, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's & Children's Hospital, Singapore
- Seoul National University Bundang Hospital, Seongnam, South Korea
- Gregorio Marañón General University Hospital, Madrid, Spain
- National Taiwan University Hospital, Taipei, Taiwan
- King Chulalongkorn University, Bangkok, Thailand
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niles DE, Duval-Arnould J, Skellett S, Knight L, Su F, Raymond TT, Sweberg T, Sen AI, Atkins DL, Friess SH, de Caen AR, Kurosawa H, Sutton RM, Wolfe H, Berg RA, Silver A, Hunt EA, Nadkarni VM; pediatric Resuscitation Quality (pediRES-Q) Collaborative Investigators. Characterization of Pediatric In-Hospital Cardiopulmonary Resuscitation Quality Metrics Across an International Resuscitation Collaborative. Pediatr Crit Care Med. 2018 May;19(5):421-432. doi: 10.1097/PCC.0000000000001520. PMID 29533355
- [Background] Sweberg T, Sen AI, Mullan PC, Cheng A, Knight L, Del Castillo J, Ikeyama T, Seshadri R, Hazinski MF, Raymond T, Niles DE, Nadkarni V, Wolfe H; pediatric resuscitation quality (pediRES-Q) collaborative investigators. Description of hot debriefings after in-hospital cardiac arrests in an international pediatric quality improvement collaborative. Resuscitation. 2018 Jul;128:181-187. doi: 10.1016/j.resuscitation.2018.05.015. Epub 2018 May 26. PMID 29768181
- [Background] Pfeiffer S, Lauridsen KG, Wenger J, Hunt EA, Haskell S, Atkins DL, Duval-Arnould JM, Knight LJ, Cheng A, Gilfoyle E, Su F, Balikai S, Skellett S, Hui MY, Niles DE, Roberts JS, Nadkarni VM, Tegtmeyer K, Dewan M; Pediatric Resuscitation Quality Collaborative Investigators. Code Team Structure and Training in the Pediatric Resuscitation Quality International Collaborative. Pediatr Emerg Care. 2021 Aug 1;37(8):e431-e435. doi: 10.1097/PEC.0000000000001748. PMID 31045955
- [Background] Esangbedo I, Yu P, Raymond T, Niles DE, Hanna R, Zhang X, Wolfe H, Griffis H, Nadkarni V; Pediatric Resuscitation Quality (pediRES-Q) Collaborative Investigators. Pediatric in-hospital CPR quality at night and on weekends. Resuscitation. 2020 Jan 1;146:56-63. doi: 10.1016/j.resuscitation.2019.10.039. Epub 2019 Nov 14. PMID 31734222
- [Background] Wolfe HA, Wenger J, Sutton R, Seshadri R, Niles DE, Nadkarni V, Duval-Arnould J, Sen AI, Cheng A. Cold Debriefings after In-hospital Cardiac Arrest in an International Pediatric Resuscitation Quality Improvement Collaborative. Pediatr Qual Saf. 2020 Jul 8;5(4):e319. doi: 10.1097/pq9.0000000000000319. eCollection 2020 Jul-Aug. PMID 32766493
- [Derived] Raymond TT, Esangbedo ID, Rajapreyar P, Je S, Zhang X, Griffis HM, Wakeham MK, Petersen TL, Kirschen MP, Topjian AA, Lasa JJ, Francoeur CI, Nadkarni VM; pediatric Resuscitation Quality (pediRES-Q) Collaborative Investigators. Cerebral Oximetry During Pediatric In-Hospital Cardiac Arrest: A Multicenter Study of Survival and Neurologic Outcome. Crit Care Med. 2024 May 1;52(5):775-785. doi: 10.1097/CCM.0000000000006186. Epub 2024 Jan 5. PMID 38180092
- [Derived] Ong GY, Chen ZJ, Niles DE, Srinivasan V, Sen AI, Skellett S, Ikeyama T, Del Castillo J, Berg RA, Nadkarni VM. Poor Concordance of One-Third Anterior-Posterior Chest Diameter Measurements With Absolute Age-Specific Chest Compression Depth Targets in Pediatric Cardiac Arrest Patients. J Am Heart Assoc. 2023 Jul 18;12(14):e028418. doi: 10.1161/JAHA.122.028418. Epub 2023 Jul 8. PMID 37421276
- [Derived] Gray JM, Raymond TT, Atkins DL, Tegtmeyer K, Niles DE, Nadkarni VM, Pandit SV, Dewan M; pediRES-Q Investigators. Inappropriate Shock Delivery Is Common During Pediatric In-Hospital Cardiac Arrest. Pediatr Crit Care Med. 2023 Aug 1;24(8):e390-e396. doi: 10.1097/PCC.0000000000003241. Epub 2023 Apr 28. PMID 37115167
- [Derived] Raymond TT, Pandit SV, Griffis H, Zhang X, Hanna R, Niles DE, Silver A, Lasa JJ, Haskell SE, Atkins DL, Nadkarni VM; Pediatric Resuscitation Quality Collaborative (pediRES-Q) Investigators. Effect of Amplitude Spectral Area on Termination of Fibrillation and Outcomes in Pediatric Cardiac Arrest. J Am Heart Assoc. 2021 Jun 15;10(12):e020353. doi: 10.1161/JAHA.120.020353. Epub 2021 Jun 5. PMID 34096341
- See also: Learn more about the platform! — https://www.pedires-q.org